CLINICAL TRIAL: NCT01697657
Title: A Randomised, Open Label, Cross-over, Multi-centre, Multinational Trial Comparing the Frequency of Hypoglycaemic Episodes During Treatment With Insulin Detemir and NPH Insulin in Well Controlled Subjects With Type 1 Diabetes on a Basal-bolus Regimen
Brief Title: Frequency of Hypoglycaemic Episodes During Treatment With Insulin Detemir in Well Controlled Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1375
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Detemir (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- NPH (Active Comparator)
  Interventions: Drug: insulin NPH; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Subjects were dosed according to individual requirements. Injected subcutaneously (s.c. under the skin) twice daily in the morning and at bedtime for 10 weeks after an initial 6-week titration in treatment period 1 followed by 10 weeks after an initial 6-week titration in treatment period 2
  Arms: Detemir
Drug: insulin NPH — Subjects were dosed according to individual requirements. Injected subcutaneously (s.c. under the skin) twice daily in the morning and at bedtime for 10 weeks after an initial 6-week titration in treatment period 1 followed by 10 weeks after an initial 6-week titration in treatment period 2
  Arms: NPH
Drug: insulin aspart — Subjects were dosed according to individual requirements. Injected subcutaneously (s.c. under the skin) twice daily before meals for 10 weeks after an initial 6-week titration in treatment period 1 followed by 10 weeks after an initial 6-week titration in treatment period 2

SUMMARY:
This trial is conducted in Africa, Europe and Oceania. The aim of this trial is to investigate whether insulin detemir combined with insulin aspart compared to NPH insulin combined with insulin aspart could reduce the frequency of hypoglycaemic episodes whilst maintaining the same degree of glycaemic control subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Fasting c-peptide below lower limit of normal fasting range
* Duration of type 1 diabetes for at least 12 months
* Current treatment: Basal - bolus regimen for at least 4 months with intermediate or long-acting insulin once, twice or three times daily as basal insulin and 3-4 premeal insulin aspart or lispro injections
* HbA1c maximum 9.0% (using Biorad Variant method)
* Able and willing to perform self-monitoring of blood glucose
* Basal insulin requirement at least 30% of the total daily insulin dose
* BMI (body Mass Index) maximum 35 kg/m^2

Exclusion Criteria:

* Proliferative retinopathy or maculopathy requiring acute treatment
* Total daily insulin dose above 1.4 IU/kg/day
* Known unawareness of hypoglycaemia
* Impaired hepatic function
* Impaired renal function
* Cardiac problems
* Uncontrolled, treated/untreated hypertension
* Known or suspected allergy to trial product or related products

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2001-09; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Incidence of total self-recorded hypoglycaemic episodes

SECONDARY OUTCOMES:
Incidence of total major hypoglycaemic episodes
HbA1c (glycosylated haemoglobin)
8-point plasma glucose profiles
Serum glucose profiles
72-hours glucose profile
Within-subject variation in home-measured fasting plasma glucose
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (11):
- Australia (3):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Ashford
  - Novo Nordisk Investigational Site, Box Hill
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Denmark (2):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Køge
- Italy (2):
  - Novo Nordisk Investigational Site, Città di Castello
  - Novo Nordisk Investigational Site, Perugia
- Novo Nordisk Investigational Site, Cape Town, Western Cape, South Africa
- Sweden (2):
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Trelleborg

REFERENCES:
- [Result] Kolendorf K, Ross GP, Pavlic-Renar I, Perriello G, Philotheou A, Jendle J, Gall MA, Heller SR. Insulin detemir lowers the risk of hypoglycaemia and provides more consistent plasma glucose levels compared with NPH insulin in Type 1 diabetes. Diabet Med. 2006 Jul;23(7):729-35. doi: 10.1111/j.1464-5491.2006.01862.x. PMID 16842476
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com